CLINICAL TRIAL: NCT04487041
Title: Tfh Dysfunction in HIV and Aging
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Savita Pahwa, Professor, University of Miami
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 20200752
Record Dates: First submitted 2020-07-22; First posted 2020-07-27 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Human Influenza
Keywords: HIV; Aging; flu vaccination; high dose vaccination; immune function
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Young HIV negative group (Active Comparator): HIV uninfected participants that are 18-35 years of age will receive the standard dose flu vaccine. Participants who did not respond to the standard dose flu vaccination, as defined by less than a four-fold increase in flu antibody titer from baseline, will then receive the high dose flu vaccination 1 year after initial standard dose flu vaccination. Participants who respond to the standard dose flu vaccination will not receive the high dose flu vaccination.
  Interventions: Biological: Standard dose influenza vaccination; Biological: High dose influenza vaccination
- Young HIV positive group (Experimental): HIV infected viral suppressed participants, who are on anti-retroviral therapy (ART) aged 18-35 years of age, will receive the standard dose flu vaccine first followed by the high dose flu vaccine 1 year after initial standard dose.
  Interventions: Biological: Standard dose influenza vaccination; Biological: High dose influenza vaccination
- Old HIV negative group (Experimental): HIV uninfected participants that are 65 years and older will receive the standard dose flu vaccine first followed by the high dose flu vaccine 1 year after initial standard dose.
  Interventions: Biological: Standard dose influenza vaccination; Biological: High dose influenza vaccination
- Old HIV positive group (Experimental): HIV infected viral suppressed participants, who are on anti-retroviral therapy (ART) aged 65 years and older, will receive the standard dose flu vaccine first followed by the high dose flu vaccine 1 year after initial standard dose.
  Interventions: Biological: Standard dose influenza vaccination; Biological: High dose influenza vaccination

INTERVENTIONS:
Biological: Standard dose influenza vaccination — Single 0.5 ml injection administered intramuscularly into participant's deltoid muscle
  Other Names: Fluzone quadrivalent
Biological: High dose influenza vaccination — 4 times more concentrated single 0.7 ml injection administered intramuscularly into participant's deltoid muscle
  Other Names: Fluzone high dose quadrivalent

SUMMARY:
The purpose of this research is to evaluate blood samples from HIV infected and non-HIV infected people to understand how aging and HIV infection affect the immune responses (body defenses against infection) to the flu vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. For HIV positive participants:

   * HIV infection, as documented by any licensed ELISA test kit. Participants on ART as a result of prior HIV documented infection will not be required to provide proof of diagnosis of HIV infection.
   * Additional criteria for HIV positive

     1. on ART for at least 1 year. Occasional viral blips up to 1000 copies/ml also acceptable provided the patients are on continuing treatment,
     2. Cluster of differentiation 4 (CD4) count available in the prior 6 months and >200/mm3
     3. Undetectable viral load (< 40 copies/mL). Blips of <1000 copies/mL will be allowed.
2. For HIV negative participants:

   * Documented negative HIV test at the time of study entry, either by any licensed ELISA.
3. For all participants:

   1. Individuals age: ≤35 years and ≥65 years.
   2. No history of other immunodeficiency disorders
   3. Not on steroid or other immunosuppressive/immunomodulators medications.
   4. No active malignancies.
   5. Agreeable to receive both regular standard (STD-TIV) and high dose (HD-TIV) influenza vaccination.
   6. Agreeable to participate in study for a complete course of study full visits including 2 consecutive flu seasons.
   7. Able to provide informed consent.

Exclusion criteria

1. Contraindication to receive influenza vaccination.
2. Non-adherence to ART for HIV positive
3. Unable to provide informed consent.
4. Influenza vaccination already given during the current vaccination season.
5. Known drug abuse including cocaine by history

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-10-30 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in HAI antibody response | Baseline to Month 6 (post standard dose flu vaccination), Baseline to Month 18 (post high-dose flu vaccination)
  Change in mean titers of Hemagglutination inhibition (HAI) antibody response will be measured using serum sample.
Change in neutralization antibody response | Baseline to Month 6 (post standard dose flu vaccination), Baseline to Month 18 (post high-dose flu vaccination)
  Change in mean titers of neutralization antibody response will be measured using serum sample.
Percentage of Participants with Vaccine Response | Month 13 (1 month post high-dose flu vaccination)
  Percentage of participants that are vaccine responders and non-responders will be reported. Response is evaluated using seroconversion to the flu vaccine using serum sample.

SECONDARY OUTCOMES:
Percentage of T-follicular helper (Tfh) cells | Month 13 (1 month post high-dose flu vaccination)
  Percentage of Tfh cells as measured using peripheral blood samples
Percentage of B cells | Month 13 (1 month post high-dose flu vaccination)
  Percentage of B cells as measured using peripheral blood samples
Percentage of monocytes | Month 13 (1 month post high-dose flu vaccination)
  Percentage of monocytes as measured using peripheral blood samples
Percentage of Tfh cells producing cytokines | Month 13 (1 month post high-dose flu vaccination)
  Percentage of Tfh cells producing cytokines as measured using peripheral blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Savita Pahwa, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No